CLINICAL TRIAL: NCT07311642
Title: The Effect of Intraoperative Binaural Beats on Remimazolam Dose Required for Maintenance of General Anesthesia: a Randomized, Placebo-controlled Trial
Brief Title: The Effect of Intraoperative Binaural Beats on Remimazolam Dose Required for Maintenance of General Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Hwa Seo, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2510-082-1686
Record Dates: First submitted 2025-12-04; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-11

CONDITIONS: Breast Reconstruction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- biaural beat (Experimental): Participants receive binaural beats via earphones from OR entry until end of surgery.
  Interventions: Device: biaural beat
- control (Active Comparator): Participants wear identical earphones but receive no audio stimulation.
  Interventions: Device: control

INTERVENTIONS:
Device: biaural beat — Participants receive binaural beats via earphones from OR entry until end of surgery.
  Arms: biaural beat
Device: control — Participants wear identical earphones but receive no audio stimulation.
  Arms: control

SUMMARY:
This prospective randomized controlled trial evaluates whether intraoperative binaural beats reduce the remimazolam dose required for general anesthesia in 88 adults undergoing breast surgery. Patients are assigned to binaural beats or silent earphones, and the primary outcome is total intraoperative remimazolam consumption.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥19 years old) scheduled to undergo breast surgery with reconstruction under general anesthesia.

Exclusion Criteria:

* Patients with hearing impairment, hearing loss, or those using hearing aids
* Patients with external auditory canal disease that prevents wearing earphones
* Patients with chronic use of hypnotics or sedatives
* Patients with a history of obstructive sleep apnea or a BMI ≥ 35 kg/m²
* Patients with alcohol dependence or substance abuse
* Patients deemed inappropriate for study participation at the discretion of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Total intraoperative remimazolam dose | From induction of anesthesia to end of surgery
  Total amount of remimazolam administered during general anesthesia

SECONDARY OUTCOMES:
Total intraoperative remifentanil dose | Intraoperative period
  Total remifentanil administered using target-controlled infusion.
BIS | Intraoperative period
  BIS levels measured continuously.
Postoperative analgesic use | PACU until Postoperative day 1
  Amount of opioids, non-opioid analgesics administered.
Heart rate | intraoperative
  Heart rate during operation
blood pressure | intraoperative
  blood pressure during surgery
SpO₂ | intraoperative
  saturation during surgery
Postoperative antiemetic use | PACU until Postoperative day 1
  Amount of antiemetics administered.